CLINICAL TRIAL: NCT07213310
Title: A Phase 1, Open-label, Fixed-sequence, Drug-drug Interaction Study to Evaluate the Effect of DWC202511 or DWC202512 on the Pharmacokinetics of DWP16001 and Its Metabolite in Healthy Adult Subjects
Brief Title: Drug-Drug Interaction Study to Evaluate the Effect of DWC202511 or DWC202512 With DWP16001 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001113
Record Dates: First submitted 2025-07-29; First posted 2025-10-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy
MeSH Terms: interventions — Enavogliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm: Sequential administration of DWC202511, DWC202512, and DWP16001 (Experimental)
  Interventions: Drug: DWP16001; Drug: DWC202511; Drug: DWC202512

INTERVENTIONS:
Drug: DWP16001 — DWP16001 enavogliflozin (single oral dose) is administered in accordance with the study protocol.
Drug: DWC202511 — Repeated oral administration of DWC202511 500 mg twice daily (BID), in accordance with the study protocol.
Drug: DWC202512 — Repeated oral administration of DWC202512 once daily, in accordance with the study protocol

SUMMARY:
Drug-Drug Interaction Study to Evaluate the Effect of DWC202511 or DWC202512 With DWP16001 in Healthy Adults

DETAILED DESCRIPTION:
A phase 1, open-label, fixed-sequence, drug-drug interaction study to evaluate the effect of DWC202511 or DWC202512 on the pharmacokinetics of DWP16001 and its metabolite in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged 19 to 50 years at the time of screening.
* 50.0 kg ≤ Body weight ≤ 90.0 kg and 18.5 ≤ Body Mass Index (BMI) ≤ 29.9 kg/m² at the time of screening.
* Written consent on voluntary decision of participation prior to the screening procedure after being fully informed of and completely understanding this study, etc.

Exclusion Criteria:

* Currect or history of clinically significant hepatic, renal, kidney, nervous, immune, respiratory, gastrointestinal, endocrine, hematologic/oncologic conditions, cardiovascular, genitourinary, psychiatric, or sexual disorders.
* History of gastrointestinal diseases (e.g., Crohn's disease, ulcers, gastritis, gastric spasms, gastroesophageal reflux disease) or surgeries (excluding simple appendectomy or hernia repair) that may affect the safety, pharmacokinetics, or pharmacodynamics of the investigational product.
* Current or history of gastrointestinal disorders or prior gastrointestinal surgery (except appendectomy or hernia repair) that may affect safety or PK/PD assessment of the investigational product.

Current or history of urinary tract infection or genital fungal infection.

* Current or history of metabolic acidosis, such as diabetic ketoacidosis.
* Genetic disorders including galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-11-09 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Cmax | 1 week
AUClast | 1 week

SECONDARY OUTCOMES:
AUCinf | 1 week
  AUCinf of DWP16001 and DWP16001 metabolites
t1/2 | 1 week
  t1/2 of DWP16001 and DWP16001 metabolites
Tmax | 1 week
  Tmax of DWP16001 and DWP16001 metabolites
CL/F | 1 week
  CL/F of DWP16001
Vz/F | 1 week
  Vz/F of DWP16001
metabolic ratio | 1 week
  metabolic ratio of DWP16001 metabolites

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jong No Gu, South Korea